CLINICAL TRIAL: NCT02278887
Title: Randomized Phase III Study Comparing a Non-myeloablative Lymphocyte Depleting Regimen of Chemotherapy Followed by Infusion of Tumor Infiltrating Lymphocytes and Interleukin-2 to Standard Ipilimumab Treatment in Metastatic Melanoma
Brief Title: Study Comparing TIL to Standard Ipilimumab in Patients With Metastatic Melanoma
Acronym: TIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14TIL
Record Dates: First submitted 2014-06-03; First posted 2014-10-30 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; TIL treatment; tumor infiltrating lymphocytes; ipilimumab; interleukin 2; non-myeloablative; randomization
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection; Cyclophosphamide; Drug Therapy; fludarabine; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab (Active Comparator): 4 cycles of ipilimumab treatment, the standard treatment
  Interventions: Procedure: Translational research; Drug: Ipilimumab infusion
- TIL treatment (Experimental): non-myeloablative lymphocyte depleting regimen of chemotherapy followed by infusion of tumor infiltrating lymphocytes and interleukin-2
  Interventions: Procedure: Translational research; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2

INTERVENTIONS:
Procedure: Translational research — Before during and at progression/regression biopsies and blood will be taken for translational research
  Other Names: tumor tissue; blood
Drug: Cyclophosphamide — The patient receives 2 days cyclophosphamide via IV to deplete T-cells.
  Other Names: chemotherapy
  Arms: TIL treatment
Drug: Fludarabine — The patient receives 5 days fludarabine via IV to deplete T-cells.
  Other Names: chemotherapy
  Arms: TIL treatment
Drug: Interleukin-2 — After infusion of the TIL, the patient receives IL-2 to keep the TIL active.
  Other Names: Proleukin
  Arms: TIL treatment
Drug: Ipilimumab infusion — In arm A patients will be treated with 4 infusion of ipilimumab
  Other Names: standard treatment
  Arms: Ipilimumab

SUMMARY:
In this randomized controlled phase III study the investigators will evaluate whether TIL infusion preceded by non-myeloablative chemotherapy and followed by high dose bolus interleukin-2 can result in an improved progression free survival when randomly compared to ipilimumab in 168 stage IV melanoma patients. A health technology assessment (HTA) will be performed to evaluate the impact of the TIL treatment on patients and organizational processes and cost-effectivity.

DETAILED DESCRIPTION:
In this randomized controlled phase III study the investigators will evaluate whether TIL infusion preceded by non-myeloablative chemotherapy and followed by high dose bolus interleukin-2 can result in an improved progression free survival when randomly compared to ipilimumab in 168 stage IV melanoma patients. A health technology assessment (HTA) will be performed to evaluate the impact of the TIL treatment on patients and organizational processes and cost-effectivity. This will be done via questionnaires at baseline, just after treatment and during follow-up. Also healthcare providers will be interviewed after 6 months after starting the trial.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable AJCC stage III or stage IV melanoma
* Patients must have metastatic melanoma with a resectable metastatic lesion(s) of sufficient size (≥ 2-3 cm in total) and must be willing to undergo such a resection for experimental purposes.
* Patients should have received maximum one line of systemic therapy (except for ipilimumab) for unresectable or metastatic melanoma.[
* Patients must be ≥ 18 years and ≤ 75 years of age and must have measurable disease by CT or MRI per RECIST 1.1 criteria (in addition to the resected lesion).
* Patients must have a clinical performance status of ECOG 0 or 1.
* Patients of both genders must be willing to practice a highly effective method of birth control during treatment and for four months after receiving the preparative regimen.
* Patients must be able to understand and sign the Informed Consent document.

Exclusion Criteria:

* Life expectancy of less than three months.
* Patients with metastatic ocular/ mucosal or other non-cutaneous melanoma.
* Adjuvant treatment with ipilimumab within 6 months prior to randomization.
* Requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive drugs within the last 3 weeks prior to randomization.
* Patients who have a more than two CNS metastases.
* Patients who have any CNS lesion that is symptomatic, greater than 1 cm in diameter or show significant surrounding edema on MRI scan will not be eligible until they have been treated and demonstrated no clinical or radiologic CNS progression for at least 2 months.
* All patients' toxicities due to prior non-systemic treatment must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures or focal palliative radiotherapy (to non-target lesions) within the past 4 weeks, as long as all toxicities have recovered to grade 1 or less.
* Women who are pregnant or breastfeeding, because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Any active systemic infections, coagulation disorders or other active major medical illnesses.
* Any autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years
  Progression free survival according to RECIST 1.1

SECONDARY OUTCOMES:
Immune related progression free survival | 3 years

OTHER OUTCOMES:
Safety | 3 years
  Adverse events will be assessed during treatment and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: John B.A.G. Haanen, Prof., Principal Investigator — The Netherlands Cancer Institute
Locations (2):
- CCIT Department of Oncology and Haematology Herlev Hospital, Copenhagen, Denmark
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Tas L, Weitemeyer MB, Rohaan MW, Borch TH, van Akkooi ACJ, Wouters MWJM, Hartemink KJ, Schrage YM, Kuijpers A, Kok NFM, van Zon M, Jedema I, Nijenhuis CM, Nuijen B, Hansen M, Voermans C, Klobuch S, Seijkens TTP, Lalezari F, Met O, Donia M, Svane IM, Haanen JBAG, Holmich LR, van Houdt WJ. Surgical considerations for tumour-infiltrating lymphocyte therapy in melanoma: results from a randomized phase III trial. Br J Surg. 2025 May 31;112(6):znaf090. doi: 10.1093/bjs/znaf090. PMID 40474841
- [Derived] Rohaan MW, Borch TH, van den Berg JH, Met O, Kessels R, Geukes Foppen MH, Stoltenborg Granhoj J, Nuijen B, Nijenhuis C, Jedema I, van Zon M, Scheij S, Beijnen JH, Hansen M, Voermans C, Noringriis IM, Monberg TJ, Holmstroem RB, Wever LDV, van Dijk M, Grijpink-Ongering LG, Valkenet LHM, Torres Acosta A, Karger M, Borgers JSW, Ten Ham RMT, Retel VP, van Harten WH, Lalezari F, van Tinteren H, van der Veldt AAM, Hospers GAP, Stevense-den Boer MAM, Suijkerbuijk KPM, Aarts MJB, Piersma D, van den Eertwegh AJM, de Groot JB, Vreugdenhil G, Kapiteijn E, Boers-Sonderen MJ, Fiets WE, van den Berkmortel FWPJ, Ellebaek E, Holmich LR, van Akkooi ACJ, van Houdt WJ, Wouters MWJM, van Thienen JV, Blank CU, Meerveld-Eggink A, Klobuch S, Wilgenhof S, Schumacher TN, Donia M, Svane IM, Haanen JBAG. Tumor-Infiltrating Lymphocyte Therapy or Ipilimumab in Advanced Melanoma. N Engl J Med. 2022 Dec 8;387(23):2113-2125. doi: 10.1056/NEJMoa2210233. PMID 36477031